CLINICAL TRIAL: NCT05077046
Title: Efficacy of an Ergonomic Handwriting Pen - a Monocenter Randomized Controlled Counter-balanced Trial
Brief Title: Efficacy of an Ergonomic Handwriting Pen - The AWP Pen Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences for Health Professions Upper Austria (Other)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: AWP-Pen 001
Record Dates: First submitted 2021-09-19; First posted 2021-10-13 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Muscle Fatigue
Keywords: Office Work; Handwriting Performance; Pain; Discomfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be informed that the effect of the handwriting pen design on different physiological parameters will be investigated within the study. Although participants know that they will execute the test battery twice with two different handwriting pens, they will receive no information on which of the pens will be the intervention of interest (intervention pen). To realize an efficient masking process, control pens will be exclusively created for the study. Control pens will be made of the same material and will contain cartridge. They will only differ in design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention first arm (Experimental): Due to the counter-balanced design of this study all participants will experience both an interventional and a control period. Within the "intervention first arm" participants will be asked to execute the assessment trial / test battery with the intervention pen first. After a wash-out period, the participants will execute the same assessment trial / test battery with the control pen.
  Interventions: Other: Ergonomic handwriting pen
- Control first arm (Experimental): Due to the counter-balanced design of this study all participants will experience both an interventional and a control period. Within the "control first arm" participants will be asked to execute the assessment trial / test battery with the control pen first. After a wash-out period, the participants will execute the same assessment trial / test battery with the intervention pen.
  Interventions: Other: Ergonomic handwriting pen

INTERVENTIONS:
Other: Ergonomic handwriting pen — An ergonomic handwriting pen called AWP-pen designed to reduce perceived muscle fatigue, finger tip pressure and discomfort during handwriting activities.

SUMMARY:
This clinical investigation is a monocenter, prospective, randomized, controlled, counter-balanced, two-arm study investigating the effect of a novel ergonomic handwriting pen.

DETAILED DESCRIPTION:
Background:

Extended and prolonged handwriting activities can be exhausting for the writer and can lead to muscle cramps, irritations in the hand and lower arm as well as high pressures in the fingers and pain. As muscle pain in the upper extremities can affect hand writing quality, and as it is well known that high tendon activities and tissue pressures can lead to health issues, there is a need for ergonomic handwriting materials, especially for people with prolonged and extended handwriting activities (e.g. students).

Despite the high number of ergonomic handwriting pens on the market, clinical or scientific investigations for such pens are very rare. Indeed only a few studies on such pens are available, and there is little knowledge on how ergonomics can impact physiological and performance parameters. As high forces and pressures in the hand region over a long period of time can lead to health issues, a pen design targeting the reduction of grip forces and pressures was developed.

To investigate if this pen design can affect handwriting performance, perceived fatigue, pen and discomfort, the AWP pen study was developed. To follow international recommendations and to reduce potential bias as well as interpersonal variation, this study was designed as randomized controlled counter-balanced trial. The insights of this study can further help to develop novel handwriting tools and to support people with handwriting disabilities (e.g. stroke patients).

Methods:

The study consists of one assessment day / visit only. During this visit and after proving the study eligibility (inclusion / exclusion criteria), half of the study participants will randomly be allocated to one of two study groups. Depending on the group allocation participants will either execute the first assessment trial with an ergonomic (= intervention) or common (= control) handwriting pen. The randomization will be realized with opaque envelopes created by an external and independent person.

Overall participants will execute the identical assessment trial / test battery with the control and the intervention pen. Each assessment trial consists of writing speed and accuracy tasks, followed by the "Handwriting Assessment Battery for Adults" (HAB) and a fatigue task. These assessments are followed by Visual Analogue Scales and a questionnaire.

Due to the counter-balanced design and the fatigue tasks, the break between both assessment trials will take at least 20 minutes to ensure similar baseline conditions for both pens. The influence of incomplete fatigue recovery as well as practice effects will be reduced by the counter-balanced design.

The overall duration of study participation ranges between 2.5 and 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* People aged between 18 and 50 years
* People free of acute or chronical diseases limiting their handwriting capabilities (e.g. Parkinson, hand/arm amputee)
* Education level: at least high school diploma
* People using a handwriting pen > once per week
* Sufficient German language skills (min. B2 level - Questionnaire language)

Exclusion Criteria:

* People with mental disorders limiting their writing performance
* People with chronical fatigue syndrome
* People incapable of concentrating on tasks for more than 30 minutes
* Non-corrected visual disturbances

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Subjectively perceived muscle fatigue changes as determined with a Visual Analogue Scale (VAS) | 1 experimental day
  Subjects will rate their subjectively perceived muscle fatigue prior and after the test battery by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (none) to 100 (strongly pronounced) points.
  Question:
  How would you describe your current muscle fatigue in your writing hand?
Subjectively perceived discomfort as determined with a Visual Analogue Scale (VAS) | 1 experimental day
  Subjects will rate their subjectively perceived discomfort in the writing hand prior and after the test battery by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (none) to 100 (strongly pronounced) points.
  Question:
  How would you describe your current discomfort in the writing hand?

SECONDARY OUTCOMES:
Muscle pain estimated as determined with a Visual Analogue Scale (VAS) | 1 experimental day
  Subjects will rate their subjectively perceived discomfort in the writing hand prior and after the test battery by means of a Visual Analogue Scale (VAS). The VAS used for this study ranges from 0 (none) to 100 (strongly pronounced) points.
  Question:
  How would you rate the current pain in the writing hand?
Handwriting speed as determined with a maze task (accuracy based) | 1 experimental day
  Within this assessments, participants are asked to follow a predefined maze task. Overall, the same maze is used twice in different sizes to realize a progressive difficulty. In addition, as muscle fatigue can affect handling accuracy, the most difficult / accuracy maze task is to be put first in the study procedure.
  The test instruction is:
  "Cross the maze as accurately as possible without any time pressure".
  In addition to a detailed test instruction, two practice mazes have to be executed by the test subjects and supervised by a study member.
  The handling speed (time required to pass the whole maze) as well as the number of errors (lines outside the walls) will be recorded and analyzed by a study member.
Handwriting speed as determined with a maze task (speed and accuracy based) | 1 experimental day
  Within this assessments, participants are asked to follow a predefined maze task. Overall, the same maze is used three times in different sizes to realize a progressive difficulty. In addition, as muscle fatigue can affect handling accuracy, the most difficult / accuracy maze task is to be put first in the study procedure.
  The test instruction is:
  "Cross the maze as soon as possible, but do not touch the walls";
  In addition to a detailed test instruction, two practice mazes have to be executed by the test subjects and supervised by a study member.
  The handling speed (time required to pass the whole maze) as well as the number of errors (lines outside the walls) will be recorded and analyzed by a study member.
Handwriting speed as determined with a dot in cycle task | 1 experimental day
  One working speed test - named dot in cycle task - is part of the study procedure. Within this test, participants are asked to draw as many dots in a cluster of cycles as possible. This test has already been used for research, and it is characterized by a very easy design.
  The test instructions for this test are:
  "Fill in as many dots in the middle of the cycles as possible. Work as fast and accurate as possible. Work from the left to right, beginning in the upper left corner."
  Similar to the maze tasks, the dot in cycle task consist of a detailed test instruction, the test itself as well as two practice tasks. The execution of these practice tasks must be supervised by a study member to:
  * ensure that the test subject fully understood the tasks,
  * get the possibility to clarify some uncertainties when the test tasks exhibit some uncertainties,
  * reduce practice effects that will occur on the regular task.
Handwriting speed as determined with a fatigue task | 1 experimental day
  The fatigue task is a simple writing task implemented to induce muscle fatigue. Within this task the test subject is asked to copy a predefined text passage by using the corresponding study pen. As noticeable fatigue occurs only after a certain writing time and intensity, this copying process will last for 15 minutes. In addition, the test subjects are asked to copy as many words as possible within this time frame.
Positioning accuracy as determined with a maze task (accuracy based) | 1 experimental day
  Within this assessments, participants are asked to follow a predefined maze task. Overall, the same maze is used twice in different sizes to realize a progressive difficulty. In addition, as muscle fatigue can affect handling accuracy, the most difficult / accuracy maze task is to be put first in the study procedure.
  The test instruction is:
  "Cross the maze as accurately as possible without any time pressure".
  In addition to a detailed test instruction, two practice mazes have to be executed by the test subjects and supervised by a study member.
  The handling speed (time required to pass the whole maze) as well as the number of errors (lines outside the walls) will be recorded and analyzed by a study member.
Positioning accuracy as determined with a maze task (speed and accuracy based) | 1 experimental day
  Within this assessments, participants are asked to follow a predefined maze task. Overall, the same maze is used three times in different sizes to realize a progressive difficulty. In addition, as muscle fatigue can affect handling accuracy, the most difficult / accuracy maze task is to be put first in the study procedure.
  The test instruction is:
  "Cross the maze as soon as possible, but do not touch the walls";
  In addition to a detailed test instruction, two practice mazes have to be executed by the test subjects and supervised by a study member.
  The handling speed (time required to pass the whole maze) as well as the number of errors (lines outside the walls) will be recorded and analyzed by a study member.
Handwriting performance as determined with the Handwriting Assessment Battery for Adults (HAB) | 1 experimental day
  The "Handwriting Assessment Battery for Adults" is a standardized handwriting assessment exhibiting high intraclass correlations and standardized values for different cohorts. It consists of three main sections containing several items estimating:
  * Pen Control & Manipulation
  * Writing Speed
  * Writing Legibility
  For the Handwriting Assessment Battery predefined guidelines for data analysis exist.
Usability as determined with a non-standardized questionaire | 1 experimental day
  The questionnaires used in this study are non-standardized questionnaires consisting of questions with nominal (e.g. yes/no), ordinal (e.g. significantly worse, worse, identical, better, significantly better) or open answers (e.g. "Please state the pros of the product you used in this study"). They were developed to estimate the user experience and satisfaction with the product under investigation as well as its usability. Apart from the regular questions, the questionnaires include a short introduction as well as brief instructions on how to complete them.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwartz, Dr. MSc BSc, Principal Investigator — University of Applied Sciences for Health Professions Upper Austria
Locations (1):
- University of Applied Sciences for Health Professions Upper Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No